CLINICAL TRIAL: NCT07092618
Title: Effectiveness of Alternative Therapies in Maintaining Weight Loss Achieved by GLP-1 Medications Post-Cessation: A Randomized, Controlled Trial
Brief Title: Effectiveness of Alternative Therapies in Maintaining Weight Loss Achieved by GLP-1 Medications Post-Cessation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AgelessRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALRx009
Record Dates: First submitted 2024-12-18; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-05

CONDITIONS: Longevity; GLP-1; Geroscience; Aging
Keywords: Longevity; Aging; Healthy Aging; GLP-1
MeSH Terms: interventions — Metformin; Sirolimus; Naltrexone; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Metformin + LDN (Experimental): Month 1: 500mg/d MET, reduce Wegovy (or equivalent) to 1.7mg/wk or Ozempic (or equivalent) to 1.0mg/wk, add LDN 1.5mg b.i.d.
  Month 2: Increase MET to 1000mg/d, reduce Wegovy (or equivalent) to 1.0mg/wk or Ozempic (or equivalent) to 0.5mg/wk, increase LDN to 3mg b.i.d.
  Month 3: Increase MET to 1500mg/d, reduce Wegovy (or equivalent) to 0.5mg/wk or Ozempic (or equivalent) to 0.25mg/wk, increase LDN to 4.5mg b.i.d.
  Months 4-12: increase MET to 2000mg/d, stop Wegovy (or equivalent) or Ozempic (or equivalent) entirely, continue LDN 4.5mg b.i.d.
  Interventions: Drug: Metformin; Drug: Naltrexone
- Metformin (Experimental): Month 1: 500mg/d MET, reduce Wegovy (or equivalent) to 1.7mg/wk or Ozempic (or equivalent) to 1.0mg/wk
  Month 2: Increase MET to 1000mg/d, reduce Wegovy (or equivalent) to 1.0mg/wk or Ozempic (or equivalent) to 0.5mg/wk
  Month 3: Increase MET to 1500mg/d, reduce Wegovy (or equivalent) to 0.5mg/wk or Ozempic (or equivalent) to 0.25mg/wk
  Months 4-12: increase MET to 2000mg/d, stop Wegovy (or equivalent) or Ozempic (or equivalent) entirely
  Interventions: Drug: Metformin
- Metformin + Rapamycin (Experimental): Month 1: 500mg/d MET, reduce Wegovy (or equivalent) to 1.7mg/wk or Ozempic (or equivalent) to 1.0mg/wk, add 1mg/wk rapamycin
  Month 2: Increase MET to 1000mg/d, reduce Wegovy (or equivalent) to 1.0mg/wk or Ozempic (or equivalent) to 0.5mg/wk, increase rapamycin to 2mg/wk
  Month 3: Increase MET to 1500mg/d, reduce Wegovy (or equivalent) to 0.5mg/wk or Ozempic (or equivalent) to 0.25mg/wk, increase rapamycin to 4mg/wk
  Months 4-12: increase MET to 2000mg/d, stop Wegovy (or equivalent) or Ozempic (or equivalent) entirely, increase rapamycin to 6mg/wk
  Interventions: Drug: Metformin; Drug: Rapamycin
- Placebo (Vitamin C) (Placebo Comparator): Month 1: 250mg/d Vitamin C, reduce Wegovy (or equivalent) to 1.7mg/wk or Ozempic (or equivalent) to 1.0mg/wk
  Month 2: Increase Vitamin C to 500mg/d, reduce Wegovy (or equivalent) to 1.0mg/wk or Ozempic (or equivalent) to 0.5mg/wk
  Month 3: Increase Vitamin C to 750mg/d, reduce Wegovy (or equivalent) to 0.5mg/wk or Ozempic (or equivalent) to 0.25mg/wk
  Months 4-12: increase Vitamin C to 1000mg/d, stop Wegovy (or equivalent) or Ozempic (or equivalent) entirely
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: Metformin — Increasing doses from 500mg/d to 2000mg/d metformin
  Arms: Metformin; Metformin + LDN; Metformin + Rapamycin
Drug: Rapamycin — Increasing doses from 1mg/wk to 6mg/wk rapamycin
  Arms: Metformin + Rapamycin
Drug: Naltrexone — Increasing doses from 1.5mg b.i.d. to 4.5mg b.i.d. low-dose naltrexone
  Arms: Metformin + LDN
Dietary Supplement: Vitamin C — Placebo control - increasing doses from 250mg/d to 1000mg/d vitamin C (ascorbic acid)
  Arms: Placebo (Vitamin C)

SUMMARY:
The goal of this randomized, controlled trial is to evaluate the effectiveness of alternative therapies (metformin alone, with rapamycin, and with low-dose naltrexone) in maintaining weight loss in patients weaning off GLP-1 medications.

The main questions it aims to answer are:

* Whether the combination of metformin, with or without rapamycin or low-dose naltrexone, will be adequate to maintain the relative weight of individuals gradually discontinuing GLP-1 receptor agonist use.
* Whether individuals discontinuing GLP-1 receptor agonist use who instead use a combination of metformin, with or without rapamycin or low-dose naltrexone, will experience less weight regain over the course of six months post-cessation than those who do not use any alternative medications.

Researchers will compare the four groups: 1) control, 2) metformin, 3) metformin + rapamycin, and 4) metformin + low-dose naltrexone, to assess changes in the percentage of weight regain, metabolic indicators (e.g., HbA1c, lipid profile), and quality of life PROs, six months after cessation of GLP-1 therapy.

Participants will:

* Administer the assigned intervention following a dosing and administration protocol provided by the study and medical team.
* Complete a medical intake for overall health status, medical history and demographic information,
* Complete patient-reported outcomes/surveys and assessments
* Complete blood work at baseline and every 16 weeks thereafter to measure CBC, CMP, and standard health biomarker panels (e.g., cholesterol, glucose, creatinine, sodium, potassium).
* Share data from health wearables with the research team throughout the study to improve the accuracy of evaluating activity, sleep, heart rate, and other related healthspan measures.

ELIGIBILITY:
Inclusion Criteria:

* Existing AgelessRx patient
* Adults (40 - 85 years of age)
* Any sex
* Any ethnicity
* BMI ≥ 22 kg/m^2
* Have been on GLP-1s (Wegovy, Ozempic, or a compounded form of GLP-1s) for at least three months before study initiation
* Have lost at least 15 lbs during their GLP-1 use

Exclusion Criteria:

* Individuals who are denied a longevity product by the AgelessRx medical team will not be asked to participate in any product specific test(s) or questionnaire(s)
* History of bariatric surgery
* Use of weight-loss medications other than GLP-1s within the past 6 months
* Age <40 years
* Contraindications to naltrexone, metformin, or rapamycin
* Significant psychiatric illness that may affect participation
* Pregnant or breastfeeding individuals

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of metformin in maintaining GLP1-induced weight loss in participants weaning off of Ozempic or Wegovy (or compounded semaglutide equivalent) | 6 months
  Participant weight will be self-reported every 4 weeks and will be compared against baseline weight as percent departure from baseline.
  1. Individuals that maintain the relative weight over the course of six months post-GLP-1 receptor agonist cessation
  2. Individuals that have less weight gain over the course of six months post-GLP-1 receptor agonist cessation using the combinatorial therapies than those who do not
Evaluate the effectiveness of metformin + rapamycin in maintaining GLP1-induced weight loss in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Participant weight will be self-reported every 4 weeks and will be compared against baseline weight as percent departure from baseline.
Evaluate the effectiveness of metformin + LDN in maintaining GLP1-induced weight loss in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Participant weight will be self-reported every 4 weeks and will be compared against baseline weight as percent departure from baseline.

SECONDARY OUTCOMES:
Evaluate the effectiveness of metformin on perceived metabolic health status in participants weaning off of Ozempic or Wegovy (or compounded semaglutide equivalent) | 6 months
  Perceived metabolic health status will be assessed by the ISQ standardized questionnaire
Evaluate the effectiveness of metformin on biological metabolic health in participants weaning off of Ozempic or Wegovy (or compounded semaglutide equivalent) | 6 months
  Biological metabolic health will be assessed by a comprehensive metabolic blood panel, with each result reported in ng/dL and placed on a normalized scale identifying the upper and lower quartiles for healthy individuals
Evaluate the effectiveness of metformin + rapamycin on perceived metabolic health status in participants weaning off of Ozempic or Wegovy (or compounded semaglutide equivalent) | 6 months
  Perceived metabolic health status will be assessed by the ISQ standardized questionnaire
Evaluate the effectiveness of metformin + rapamycin on biological metabolic health in participants weaning off of Ozempic or Wegovy (or compounded semaglutide equivalent) | 6 months
  Biological metabolic health will be assessed by a comprehensive metabolic blood panel, with each result reported in ng/dL and placed on a normalized scale identifying the upper and lower quartiles for healthy individuals
Evaluate the effectiveness of metformin + LDN on perceived metabolic health status in participants weaning off of Ozempic or Wegovy (or compounded semaglutide equivalent) | 6 months
  Perceived metabolic health status will be assessed by the ISQ standardized questionnaire
Evaluate the effectiveness of metformin + LDN on biological metabolic health in participants weaning off of Ozempic or Wegovy (or compounded semaglutide equivalent) | 6 months
  Biological metabolic health will be assessed by a comprehensive metabolic blood panel, with each result reported in ng/dL and placed on a normalized scale identifying the upper and lower quartiles for healthy individuals
Evaluate the effectiveness of metformin on mood-related quality of life in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Quality of life will be assessed by the PANAS standardized questionnaire
Evaluate the effectiveness of metformin on physical health-related quality of life in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Quality of life will be assessed by the SF-36 standardized questionnaire
Evaluate the effectiveness of metformin + rapamycin on mood-related quality of life in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Quality of life will be assessed by the PANAS standardized questionnaire
Evaluate the effectiveness of metformin + rapamycin on physical health-related quality of life in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Quality of life will be assessed by the SF-36 standardized questionnaire
Evaluate the effectiveness of metformin + LDN on mood-related quality of life in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Quality of life will be assessed by the PANAS standardized questionnaire
Evaluate the effectiveness of metformin + LDN on physical health-related quality of life in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Quality of life will be assessed by the SF-36 standardized questionnaire
Evaluate the effectiveness of metformin on tolerability of treatment in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Tolerability of treatment will be extrapolated from an extensive medical questionnaire sent to participants monthly and recorded throughout the trial
Evaluate the effectiveness of metformin on long-term weight management practices in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Long-term weight management effectiveness will be assessed by reporting observed health changes as percent change in weight from baseline
Evaluate the side effects of metformin in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Side effects will be monitored via an extensive medical questionnaire sent to participants monthly and recorded throughout the trial
Evaluate the effectiveness of metformin + rapamycin on tolerability of treatment in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Tolerability of treatment will be extrapolated from an extensive medical questionnaire sent to participants monthly and recorded throughout the trial
Evaluate the effectiveness of metformin + rapamycin on long-term weight management practices in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Long-term weight management effectiveness will be assessed by reporting observed health changes as percent change in weight from baseline
Evaluate the side effects of metformin + rapamycin in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Side effects will be monitored via an extensive medical questionnaire sent to participants monthly and recorded throughout the trial
Evaluate the effectiveness of metformin + LDN on tolerability of treatment in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Tolerability of treatment will be extrapolated from an extensive medical questionnaire sent to participants monthly and recorded throughout the trial
Evaluate the effectiveness of metformin + LDN on long-term weight management practices in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Long-term weight management effectiveness will be assessed by reporting observed health changes as percent change in weight from baseline
Evaluate the side effects of metformin + LDN in participants weaning off of Ozempic (or equivalent) or Wegovy (or equivalent) | 6 months
  Side effects will be monitored via an extensive medical questionnaire sent to participants monthly and recorded throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Morgan, PhD, Principal Investigator — AgelessRx
Locations (1):
- AgelessRx, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: IPD will be shared with Institutional Review Board (IRB) approval or at the discretion of the PI/Sponsor